CLINICAL TRIAL: NCT02163005
Title: Gadolinium Enhanced Dual-Energy Computed Tomography: A Feasibility Study to Assess Image Quality and Diagnostic Confidence
Brief Title: A Feasibility Study to Assess the Use of Gadolinium in Computed Tomography
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No patients enrolled as study did not move to enrollment stage
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Amita Sharma, MD, Radiologist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012P002535a
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Contrast Media Allergy
Keywords: GDL contrast agent
MeSH Terms: interventions — Gadolinium; gadoterate meglumine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gadolinium enhancement (Experimental): Gadolinium enhancement will be performed using intravenous Dotarem[recommended dose of 0.2 mL/kg (0.1 mmol Gd/kg )]
  Interventions: Drug: Gadolinium

INTERVENTIONS:
Drug: Gadolinium — -agent will be administered intravenously and a CT scan will be performed to evaluate contrast enhancement characteristics of the agent to assess its feasibility as an alternative to Iodine based contrast agents.
  Other Names: Dotarem

SUMMARY:
Patients with an allergy to iodine based intravenous contrast cannot undergo a CT scan with contrast, unless they are premedicated. Premedication can result in a delay in diagnosis, that can be significant with acute conditions such as Pulmonary embolism.

The investigators are evaluating the use of Gadolinium as an alternative contrast agent in CT. Gadolinium has been used extensively in MRI exams but the dose that is used is not sufficient to provide good enhancement on CT. Dual Energy CT is a new technology that has better sensitivity to lower doses of intravenous contrast and the investigators aim to study its effectiveness in improving the enhancement with Gadolinium. The investigators will compare enhancement of Iodine with enhancement of Gadolinium during Dual Energy CT, to assess the possibility that Gadolinium could be used as an alternative for patients who are suspected of having Pulmonary embolism. They will recruit up to 50 patients who are having a routine Chest CT during treatment for a malignancy and administer Gadolinium contrast and Iodine contrast during a chest CT exam. The enhancement with the two agents can be compared.

DETAILED DESCRIPTION:
Although safe in most patients, iodine may be associated with lifethreatening adverse events, particularly in high-risk patient. This application is of particular clinical significance in patients with conditions like pulmonary embolism which could be fatal. CT pulmonary angiogram (CTPA) with sensitivity of 83-100% and specificity of 89-97% is currently the gold standard for diagnosis of pulmonary embolism. However, in patients who have allergy to iodinated contrast agent, CTPA cannot be performed. Gadolinium based contrast agent can serve as a viable alternative in such patients and can be used for Gadolinium enhanced MR pulmonary angiography (MRPA) and CTPA. Gadolinium enhanced MRPA however has inherent limitations in evaluating pulmonary embolism as evident from multicentre prospective study (PIOPED III) which reported technically inadequate exams in as many as 25% of patients (range 11% to 52%). The MRPA sensitivity was also low in the range of 78%. Moreover, unlike CT, low spatial and temporal resolution of MR hampers precise evaluation of lung parenchyma. Previously investigators have evaluated gadolinium enhanced CTPA on a single energy CT (SECT) at different tube potential (80 - 120 kV) and reported encouraging results. However, these patients received higher volume of gadolinium contrast (mean 53 ml, range 30-64 ml) and in spite, the scans performed at 120 kV demonstrated overall suboptimal pulmonary artery enhancement. These limitations can be potentially over come with dual-energy CT which simultaneously acquires low and high energy data. From this data, monochromatic images can be reconstructed at any desired energy from 40 keV to 140 keV.

The investigators aim to recruit up to 50 patients who will guide in determining gadolinium contrast volume, injection rate and image delay required to maximize pulmonary arterial enhancement.

ELIGIBILITY:
Inclusion Criteria:

* patients required to undergo a clinically indicated CT examination

Exclusion Criteria:

* subject less than 56 yrs of age
* pregnant women
* Non English speaking
* Abnormal Renal function
* Allergy to Gadolinium

Min Age: 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Vessel enhancement | Within 1 hour of contrast administration
  Following injection of Gadolinium based intravenous contrast, a CT scan will be performed and the level of enhancement of vessels by Gadolinium based contrast will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Amita Sharma, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States